CLINICAL TRIAL: NCT07268391
Title: SPEctral CT and miRna In Acute Myocardial Infarction for Comprehensive Adverse Remodeling Evaluation
Brief Title: Using Advanced CT Scans and Blood Markers to Better Understand Heart Damage and Recovery After a Heart Attack
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Biomédica de Salamanca (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SPECTRAMI-CARE; PI2025 03 1870 (Other: Ethics Committee for Clinical Research, Salamanca)
Record Dates: First submitted 2025-11-18; First posted 2025-12-05 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Acute Myocardial Infarction (AMI)
Keywords: magnetic resonance; miRNA; myocardial infarction; adverse ventricular remodeling; spectral computed tomography
MeSH Terms: conditions — Myocardial Infarction | interventions — Hematologic Tests

STUDY DESIGN:
Intervention Model Description: This is a multicenter, observational study with prospective enrollment of adult patients experiencing a first ST-segment elevation myocardial infarction (STEMI) (n = 95), according to the following inclusion criteria:
  * Hospital admission due to STEMI, treated in accordance with current clinical practice guidelines.
  * Left ventricular systolic dysfunction, defined as a left ventricular ejection fraction (LVEF) < 50%, assessed by transthoracic echocardiography (TTE) within the first 24-72 hours of admission.
  * Provision of signed informed consent.
  At the coordinating center (CAUSA), a control group (n = 20) will be included, consisting of patients with a clinical indication for cardiac CT for reasons other than myocardial infarction, meeting the following criteria: absence of myocardial injury or structural heart disease, ≤1 cardiovascular risk factor, LVEF > 55%, and no significant valvular disease (grade < III).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): At the coordinating center (CAUSA), a control group (n = 20) will be included, consisting of patients with a clinical indication for cardiac CT for reasons other than myocardial infarction, meeting the following criteria: absence of myocardial injury or structural heart disease, ≤1 cardiovascular risk factor, LVEF > 55%, and no significant valvular disease (grade < III).
  Interventions: Procedure: Blood analysis and spectral CT study
- Adult patients experiencing a first ST-segment elevation myocardial infarction (STEMI) (Experimental): Patientes will be included in this group if the following requirements are met:
  Hospital admission due to STEMI, treated in accordance with current clinical practice guidelines.
  Left ventricular systolic dysfunction, defined as a left ventricular ejection fraction (LVEF) < 50%, assessed by transthoracic echocardiography (TTE) within the first 24-72 hours of admission.
  Provision of signed informed consent.
  Interventions: Procedure: Blood analysis, spectral CT scan and cardiac magnetic resonance imaging (CMR) study

INTERVENTIONS:
Procedure: Blood analysis, spectral CT scan and cardiac magnetic resonance imaging (CMR) study — After providing informed consent, patients will undergo blood sampling, a spectral CT scan scheduled between the 3rd and 7th day of hospitalization (acute phase), and a cardiac magnetic resonance imaging (CMR) study performed within a maximum of 72 hours from the CT.
  Arms: Adult patients experiencing a first ST-segment elevation myocardial infarction (STEMI)
Procedure: Blood analysis and spectral CT study — Patients who meet the inclusion criteria for the control group will be invited to participate in the study. They will undergo blood sampling and the planned spectral CT study, including a late iodine enhancement acquisition.
  Arms: Control group

SUMMARY:
Acute myocardial infarction with ST-segment elevation (STEMI) remains a leading cause of morbidity and mortality worldwide. Although advances in reperfusion therapy have reduced early mortality, many patients later develop adverse ventricular remodeling (AVR), which increases the risk of heart failure and cardiovascular death. Current imaging methods, such as echocardiography and cardiac magnetic resonance (CMR), provide valuable prognostic information but have limitations in availability, cost, and their ability to predict AVR early and individually.

Spectral computed tomography (CT) is an emerging imaging technique that can characterize myocardial tissue, quantify infarct size, assess microvascular obstruction, and detect complications, with lower contrast and radiation requirements compared to conventional CT. In parallel, circulating microRNAs (miRNAs) have been identified as stable and non-invasive biomarkers that reflect key biological processes in post-infarction remodeling. Several miRNAs are linked to fibrosis, apoptosis, and ventricular remodeling, suggesting their potential to complement imaging findings in risk prediction.

This study proposes a multicenter, prospective cohort of patients with STEMI and reduced left ventricular function to evaluate whether combining spectral CT tissue characterization with serum miRNA profiling can improve early prediction of AVR. The main objective is to generate and validate a multiparametric prognostic model integrating imaging and molecular biomarkers to identify high-risk patients who may benefit from closer monitoring and tailored therapeutic strategies.

DETAILED DESCRIPTION:
Background and Rationale Acute myocardial infarction with ST-segment elevation (STEMI) continues to represent a major public health challenge, being one of the leading causes of morbidity and mortality worldwide. Advances in reperfusion therapy, particularly primary percutaneous coronary intervention (PCI), have substantially reduced short-term mortality rates. Nevertheless, a large proportion of patients experience adverse ventricular remodeling (AVR) during follow-up. AVR is characterized by pathological changes in left ventricular (LV) geometry, wall thinning, chamber dilation, and progressive decline in contractile function. These changes are strongly associated with the development of heart failure and increased long-term mortality.

Traditional imaging modalities, such as echocardiography and cardiac magnetic resonance (CMR), have been used to characterize post-infarction myocardial damage and to monitor remodeling. Echocardiography is widely available and provides important functional information, but it lacks the ability to characterize myocardial tissue in depth. CMR is currently the gold standard for infarct size quantification, detection of microvascular obstruction, and assessment of myocardial viability; however, it is costly, time-consuming, and not universally accessible. There remains an unmet need for more accessible, rapid, and accurate tools to predict AVR early after STEMI.

Spectral computed tomography (CT) has recently emerged as an innovative imaging technique that goes beyond conventional CT by providing spectral information and material decomposition. This technology enables enhanced tissue characterization, accurate quantification of myocardial perfusion defects, and identification of complications such as myocardial rupture or thrombus, all while using reduced contrast volume and lower radiation doses compared with older-generation scanners. Preliminary data suggest that spectral CT can approximate some of the information traditionally obtained through CMR, potentially offering a more accessible tool for post-infarction risk stratification.

In parallel, circulating microRNAs (miRNAs) have been identified as highly stable, non-invasive biomarkers involved in key biological processes relevant to cardiac remodeling, including fibrosis, apoptosis, angiogenesis, and inflammatory signaling. Several miRNAs have been associated with infarct size, LV dysfunction, and clinical outcomes in patients with acute myocardial infarction. Integrating molecular biomarkers with imaging could provide a powerful multiparametric model for early prediction of AVR, guiding patient-tailored therapeutic strategies.

The SPECTRAMI-CARE study (SPEctral CT and miRna In Acute Myocardial Infarction for Comprehensive Adverse Remodeling Evaluation) is designed as a prospective, multicenter observational cohort. The protocol aims to evaluate the complementary role of spectral CT and circulating miRNAs in predicting adverse remodeling after STEMI with impaired LV function.

Imaging Procedures

Spectral CT:

Performed within the first week after STEMI. Parameters include assessment of infarct size, perfusion defects, myocardial edema, and complications (e.g., thrombus, aneurysm). Quantitative indices will be derived from material decomposition images, iodine density maps, and virtual monoenergetic reconstructions.

Cardiac MRI (sub-cohort):

Used as a reference standard for infarct size, microvascular obstruction, and myocardial viability. Data will be compared with spectral CT findings for concordance and accuracy.

Echocardiography:

Performed at baseline and follow-up for routine functional assessment (LV volumes, LVEF, diastolic function, right ventricular parameters).

Molecular Biomarker Assessment Peripheral blood samples will be collected at baseline (≤72h after PCI), at 1 month, and at 3 months. miRNA profiling will be performed using next-generation sequencing and validated with quantitative RT-PCR. Candidate miRNAs previously implicated in fibrosis, apoptosis, angiogenesis, and remodeling will be specifically analyzed. Expression levels will be correlated with imaging findings and clinical outcomes.

Statistical Analysis Sample size will be based on expected incidence of AVR (~30% in high-risk STEMI populations). Multivariable logistic regression and Cox proportional hazards models will be used to identify predictors of AVR and clinical outcomes. Model performance will be evaluated using C-statistics, calibration plots, and net reclassification improvement (NRI). Internal validation will be performed with bootstrapping; external validation will be explored in an independent cohort.

Ethics and Dissemination The study will comply with the Declaration of Helsinki and local ethics regulations. Informed consent will be obtained from all participants. Data will be anonymized and stored securely. Results will be disseminated through peer-reviewed publications and presentations at scientific conferences, with the aim of contributing to precision medicine in post-infarction care.

Significance SPECTRAMI-CARE is expected to provide novel insights into the early identification of patients at risk for adverse remodeling after STEMI. By integrating cutting-edge imaging and molecular biomarkers, this study seeks to advance risk stratification and facilitate personalized strategies to improve outcomes. Spectral CT, if validated against CMR, may offer a more accessible alternative for myocardial tissue characterization, while circulating miRNAs may add a non-invasive layer of biological information. The multiparametric model proposed has the potential to change clinical practice by identifying high-risk patients earlier and enabling targeted therapeutic interventions.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years.
* First STEMI treated with primary PCI.
* Left ventricular ejection fraction (LVEF) ≤45% during index hospitalization.
* Ability to provide informed consent.

Exclusion Criteria:

* Contraindication to iodinated contrast media.
* Chronic kidney disease with eGFR <30 mL/min/1.73 m².
* Prior myocardial infarction or known cardiomyopathy.
* Contraindication to CT or MRI imaging.
* Life expectancy <1 year due to non-cardiac conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse ventricular remodeling at 6 months, defined as an increase in LV end-diastolic volume ≥20% compared with baseline. | 6 months
  The primary endpoint will be the occurrence of adverse ventricular remodeling (AVR) as assessed by cardiac magnetic resonance imaging (CMR). AVR will be defined as an increase in left ventricular end-diastolic volume (LVEDV) of ≥20% compared with baseline values obtained during the acute phase (3-7 days post-STEMI). In cases where CMR is not feasible, spectral CT-derived LV volumes will be used as a contingency reference, given their validated correlation with CMR measurements.

SECONDARY OUTCOMES:
Infarct size characterization by spectral CT vs. CMR. | Baseline and 6 months
  Quantitative assessment of infarct size will be performed using spectral CT (late iodine enhancement, iodine concentration maps, and non-contrast acquisitions for edema) and compared with CMR (late gadolinium enhancement, T1/T2 mapping, and extracellular volume fraction).
Myocardial characterization by spectral CT vs. CMR. | Baseline and 6 months
  Quantitative assessment of myocardial markers such as microvascular obstruction (MVO), intramyocardial hemorrhage, and myocardial edema will be evaluated to determine the diagnostic accuracy and reproducibility of spectral CT (late iodine enhancement, iodine concentration maps, and non-contrast acquisitions for edema) and compared with the gold standard CMR (late gadolinium enhancement, T1/T2 mapping, and extracellular volume fraction).
Correlation of miRNA signatures with remodeling. | Baseline and 6 months
  Serum miRNA profiles obtained at baseline (acute phase) and at 6 months will be analyzed to identify differential expression patterns associated with adverse remodeling.
  Specific miRNAs previously linked to fibrosis, apoptosis, and inflammation (e.g., miR-1, miR-21, miR-30a-5p, miR-133a, miR-210-3p, miR-221-3p) will be quantified by RT-qPCR.
  Qualitative correlation between miRNA expression levels and imaging-defined markers of remodeling will be tested, including potential sex-specific differences.
Predictive accuracy of integrated models (spectral CT + miRNA vs. conventional predictors) | 6 months
  Predictive models will be developed combining spectral CT-derived parameters, miRNA signatures, and conventional clinical predictors (age, sex, infarct location, Killip class, biomarkers).
  Model performance will be assessed using machine learning approaches (logistic regression, random forest, XGBoost), with internal validation through repeated 10-fold cross-validation.
  Predictive accuracy will be reported using receiver-operating characteristic (ROC) curves, area under the curve (AUC), calibration statistics, and Shapley values for interpretability.
  All parameters sill be used simultaneously to predict integrated models, therefore they cannot be sepparated in different outcomes.
Major adverse cardiovascular events (MACE) | From baseline to 6 months
  The composite endpoint of MACE will include cardiovascular death, recurrent myocardial infarction, and hospitalization for heart failure during the 12-month follow-up period.
  All events will be adjudicated by an independent clinical events committee, blinded to imaging and biomarker results.
Safety outcomes: incidence of contrast-induced nephropathy | From baseline to 6 months
  Safety outcomes will be carefully annotated, including incidence of contrast-induced nephropathy (defined as a ≥30% decline in estimated glomerular filtration rate compared with baseline).
Safety outcomes: allergic or hypersensitivity reactions | From baseline to 6 months
  Aallergic or hypersensitivity reactions to iodinated contrast or gadolinium-based agents will be assessed.
Safety outcomes: arrhythmias related to imaging procedures | From baseline to 6 months
  Arrhythmias temporally related to imaging procedures (e.g., during CT or CMR acquisition) will be evaluated.
Safety outcomes: Cumulative radiation exposure | From baseline to 6 months
  Cumulative radiation exposure from spectral CT will also be recorded and reported as an additional safety metric.

CONTACTS AND LOCATIONS:
Locations (5):
- Spain (5):
  - Centro Nacional de Investigaciones Cardiovasculares (CNIC), Madrid
  - Hospital La Princesa, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Complejo Asistencial Universitario de Salamanca, Salamanca
  - Hospital Clínico Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Plan Description: De-identified individual participant-level data (IPD) will be shared, including:
  Demographic and clinical variables collected in REDCap. Quantitative spectral CT parameters (iodine maps, first-pass perfusion, late iodine enhancement, volumetric data).
  Cardiac MRI parameters (volumes, T1/T2 mapping, ECV, MVO, IMH). Serum miRNA panel results (derived files and processed tables). Clinical outcomes (adverse ventricular remodeling defined by indexed EDV/ESV, 1-year MACE, renal function, etc.).
  Supporting documents (data dictionary, eCRFs, analysis scripts in R/Python when available, FAIR metadata) will also be provided.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Beginning 12 months after publication of primary results, available for at least 5 years.
Access Criteria: Access Criteria: Access will be granted to qualified researchers with a methodologically sound proposal. Requests will be reviewed by the study Data Committee/steering committee. Applications must be addressed to the PI (Candelas Pérez del Villar). Requirements include: Data Use Agreement (DUA), commitment to non-reidentification, appropriate data security, mandatory citation of dataset source and DOI. Analytical code sharing and a publication plan may be required prior to access approval.
  IPD Sharing Support: Data will be hosted on controlled project infrastructure (XNAT/Core-lab) and disseminated through the IBSAL Zenodo community with DOI and regulated access, in compliance with GDPR/LOPDGDD and CEIm approval.